CLINICAL TRIAL: NCT06534177
Title: Development of Digital Diagnostics and Intervention Services for Parkinson's Disease
Brief Title: Digital Diagnostics and Intervention Services for Parkinson's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: University of Exeter (Other)
Collaborators: GaitQ company (Unknown)
Responsible Party: Sponsor
Other Study IDs: 340549
Record Dates: First submitted 2024-07-29; First posted 2024-08-02 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Joint Diseases; Musculoskeletal Diseases; Parkinson Disease; Basal Ganglia Diseases; Movement Disorders; Synucleinopathies; Neuro-Degenerative Disease; Demyelinating Disease, Autoimmune, CNS; Demyelinating Disease; Autoimmune Diseases; Immune System Diseases; Bone Diseases, Metabolic; Bone Diseases; Arthritis; Osteoporosis; Multiple Sclerosis
Keywords: parkinson's disease; osteoarthritis; stroke; MS; osteoporosis
MeSH Terms: conditions — Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Joint Diseases; Musculoskeletal Diseases; Parkinson Disease; Basal Ganglia Diseases; Movement Disorders; Synucleinopathies; Demyelinating Autoimmune Diseases, CNS; Demyelinating Diseases; Autoimmune Diseases; Immune System Diseases; Bone Diseases, Metabolic; Bone Diseases; Arthritis; Osteoporosis; Multiple Sclerosis; Osteoarthritis; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with long-term conditions affecting movement: A total number of 50 people with long-term conditions affecting their movement include people with Parkinson's
- Healthy control: A total number of 30 healthy people with no condition impacting their movement and walking ability.

SUMMARY:
People with Parkinson's have infrequent clinical consultation (once every 12-18 months) and limited rehabilitation.

Assessment play an important role in these consultations to help clinicians understand patients' health status and disease progression necessary to adjust treatment plans. The current way of measuring is the UPDRS which needs a clinician to do this and takes 30 minutes. There is a strong need for more frequent and accurate Parkinson's assessments in the clinic and at home to detect changes early and then give appropriate support and drug and physiotherapy quickly. There is a need to develop good home digital physiotherapy tools to increase the amount of therapy. Here the investigators are testing new digital technologies to do these assessments in the home and clinic and a new digital physiotherapy device in the home. The investigators aim to conduct a clinical study with 50 people with Parkinson's (50 from UK) with the UPDRS, (a rating scale that is commonly used in clinical settings to evaluate the progression of Parkinson's disease) and 30 healthy adults. The investigators will develop and investigate if two new digital devices, one the MachineMD that measures eye movement and one the gaitQ that measures gait can be used instead of the MDS-UPDRS (motor) using digital gait and ophthalmic features in the clinic setting. The investigators will investigate the effect of a physiotherapy gait intervention gaitQ Tempo in the home context for two weeks and of doing the gait measure at home. The investigators will determine the potential of the gaitQ intervention to improve key gait metrics in order to collect clinical evidence and of using the gaitQ as a cuing system over a 2-week period on gait and other movement measures in the home and community

DETAILED DESCRIPTION:
Diagnosis: The current state of the art in diagnosing PD primarily revolves around clinical assessments based on symptomatology and neurological examination. The most widely used criteria for diagnosis are Movement Disorder Society (MDS) criteria and instrument (i.e. The MDSUPDRS). These criteria are highly dependent on the expertise of the diagnosing physician, and thus, are subject to variability. Furthermore, these clinical assessments are unable to accurately track disease progression over time, making it difficult to provide personalized care.

Assessment: plays an important role in these consultations to help clinicians understand patients' health status and disease progression necessary to adjust treatment plans. Current clinical methods rely on the UPDRS a standard clinical outcome measure that requires clinical expertise and training and is thus measured at clinical appointments.

Further information may be gained from patients' subjective description of their symptoms and/or via some short walking tests, such as 3 meter Timed Up and Go (TUG) performed as a snapshot in the clinic. However, patients' vary through and between days and subjective descriptions rely on their memory and observations at home. These recollections can be unreliable or lack enough detail (particularly when the patient has cognitive impairment). Walking tests, although quick to perform, show high variability due to natural fluctuations of the Parkinson's symptoms throughout the day, on/off medication status as well as the 'performing' effects when doing activities in a clinical setting. Consequently, Parkinson's care regimes are often provided on a trial-and-error basis, with resulting general delay in offering care, with early signs of disease progression often missed until conditions become more severe, and interventions such as physiotherapy are often provided too late. Hence, there is a strong need for more frequent and accurate Parkinson's assessments in a real-world environment to enable more targeted care and preventative measures and interventions via early detection of disease inflection points. Here the investigators propose to evaluate three digital approaches to see if they provide further information to support clinical decision making using gait and ophthalmic features. The current state-of-the-art in neurological diagnostics includes a range of traditional clinical examination techniques, such as manual neuro-ocular and neuro-motor function assessments, as well as more technologically advanced tools, such as imaging technologies (e.g., MRI) and electrophysiological tests (e.g., ECG). While these methods have undoubtedly contributed to significant advances in the detection and management of neurological disorders, they also present several limitations that digital approaches overcome. Traditional examinations of neurological function, such as manual assessments [UPDRS], are heavily reliant on the expertise and subjective judgment of specialized neurologists. This leads to known inconsistencies in interpreting and scoring patient performance over time, particularly in the case of neurodegenerative diseases like Parkinson's disease (PD), where patients typically consult different resident neurologists over several years.

Additionally, manual examinations lack precise measurement instruments, resulting in a low precision of observed measurements (typically ~ 2 cm) and the inability to detect early-stage, subclinical signs. PD is a complex and progressive neurodegenerative disorder with significant variability in clinical manifestations and disease progression.

Its diagnosis and monitoring remain a challenge, primarily relying on clinical examinations that are subjective and often do not capture the full extent of symptom fluctuations.

Intervention:

Enabling independent living for an ageing society is a key challenge for the UK and other developed countries. The number of patients with LTCs are increasing and already have the greatest healthcare needs of the population, requiring 50% of all GP appointments and 70% of all bed days and their treatment and care absorbs 70% of acute and primary care budgets in England. Maintaining safe mobility is a critical factor affecing life quality and life roles and responsibilities. Considering Parkinson's alone, an analysis has shown that 1 in every 37 people will be diagnosed with PD in their lifetime (2). FOG and FSG are severely debilitating aspects of the disease which greatly reduce the quality of life of PwP and contribute to the two-fold increased fall risk and related injuries (2). It is vital that The investigators provide a solution to support PwP with a more fluid and safe gait, greater independence and better disease management and care. Cueing with visual, auditory or somatosensory stimuli is a well-documented and clinically validated method to overcome FOG IRAS Form Reference: IRAS Version 6.3.6

Date:

8 340549/1665763/37/423 and FSG. Research studies have also shown that cueing modalities improve gait in PwP during both free and treadmill walking, whilst improving balance and reducing the need for stabilising support. Gait parameters such as step frequency, stride length and gait symmetry, have been shown to be measurable with inertial motion sensors for gait quality assessment. Studies have shown that objective measurement of the disease can improve treatment outcomes in PD. There are basic visual and rhythmic cueing products available (such as laser shoes, a metronome app and a vibrational button), however they are still based on simple continuous cues which have profound limitations on usability and effectiveness in the everyday environment and do not include gait analytics systems to facilitate better patient outcome and experience. The gaitQ system will be the first unique solution that uses artificial intelligence and smart adaptive cueing to help patients effectively overcome FOG and FSG in their daily environment while improving gait quality. A prior proof-of-concept academic study run at the University of Oxford in 2019 prior to gaitQ company formation, evaluated responsive vibration cueing using 17 patients over 31 hours in a clinical setting. This study demonstrated that responsive cueing can reduce FOG and improve gait quality. More recently, NIHR i4i Connect funding (completed in November 2021) enabled gaitQ to advanced its research device to a commercial prototype and conduct in-house product evaluation with 22 PwP. 91% of participants reported a positive impact of the gaitQ device: it helped prompt leg movement, increase focus during walking, maintain pace, and boost confidence in walking. The quantitative analysis of gait metrics has shown around 60% reduction of FOG and FSG events in both duration and occurrence. Moreover, participants' stride length increased by 11% while step frequency decreased by 16%; both are key outcomes towards more natural and stable walking. Our machine learning algorithms have been tested against two Parkinson's studies, achieving an average of 87% sensitivity and 85% specificity. Ongoing validation in the lab is further determining the validity and reliabiity of the gait metric and estimating the effect of the cuing on transfers and mobility and enduriance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease (UK Brain Bank Criteria) or other appropriate condition specific scale [stroke, multiple sclerosis, arthritis or osteoporosis]
* Able to self-report history of daily gait freezing and/or festination for people with PD or gait and/or transfers affected by condition
* Able to walk unsupported or using an aid for at least 5 minutes and satisfactory completion of the Canadian PARQ and if over 69 used to carrying out this level of exercise
* Adult (+18 years old)
* Normal or corrected-to-normal vision (Snellen Visual Acuity > 12/18) or safe to mobilise with support
* Montreal Cognitive assessment score >21 or ability to follow 2 stage commands Healthy participants [Phase 1,2,3]
* With no long-term conditions affecting movement
* Able to walk unsupported or using an aid for at least 3 minutes and satisfactory completion of the Canadian PARQ and
* if over 69 used to carrying out this level of exercise
* Adult (+18 years old)
* Normal or corrected-to-normal vision (Snellen Visual Acuity > 12/18) or safe to mobilise with support
* Montreal Cognitive assessment score >21 or ability to follow 2 stage commands

Exclusion Criteria:

* Participants with long-term conditions affecting movement
* Any physical or mental condition affecting ability to safely participate in this level of activity and capacity to understand
* testing as demonstrated by ability to safely follow commands and pass the PARQ by the research team.
* Cognitive impairment affecting ability to safely participate and follow instructions
* Any injury or disorder that may affect balance (other than Parkinson's or referring primary condition)
* Any skin conditions or broken skin in the calf and behind knee area
* Deep brain stimulation or pacemaker implants or other implant that may interfere with the measurement system Healthy participants
* Any physical or mental condition affecting ability to safely participate in this level of activity and capacity to understand
* testing as demonstrated by ability to safely follow commands and pass the PARQ by the research team.
* Cognitive impairment affecting ability to safely participate and follow instructions
* Any injury or disorder that may affect balance (other than Parkinson's or referring primary condition)
* Any skin conditions or broken skin in the calf and behind knee area
* Deep brain stimulation or pacemaker implants or other implants that may interfere with the measurement system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruiting adult males and females, both healthy and those with neurodegenerative disease ie. Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Lab validation of MachineMD opthalamic device vs UPDRS | 2 weeks
  To determine criterion validity to the UPDRS by describing the extent of the relationship of the digital measures taken during mobility testing and neuro-Opthalmic testing in the lab/clinic to the UPDRS
Reliability testing of GaitQ wearable device | 2 weeks
  To determine the extent of the reliability of the digital measures in the context of test-retest reliability taken over 2 weeks in a lab/clinic setting
Home/community validation | 2 weeks
  To determine day to day gaitQ metrics taken during standard testing tasks of TUG, 15 m walk and 5-minute walk in the home/community setting to establish criterion validity to the lab measures and the day-to-day variability of the gaitq tempo measures to determine minimal detectable change
Home/community validation | 2 weeks
  To describe the feasibility of daily measuring in the home of gaitQ tempo to determine usability and acceptability from metrics and completion of measures
Reliability data collection for determining minimally important differnce | 2 weeks
  To determine initial values of the gaitQ of minimally important difference in relation to the TUG scores taken during the same period in the home sertting
Determine intervention potential | 2 weeks
  To determine the potential for effect of the gaitQ intervention to improve key gait metrics taken during the standard tasks of TUG, 5-minute walk and 15 m walk, in order to collect clinical evidence as determined by responsiveness, of using the gaitQ as a cuing system over a 2-week period on gait and other movement measures in the home and community